CLINICAL TRIAL: NCT01188564
Title: A Phase III Randomized, Double-blind, Placebo-controlled Study With an Open-label Extension Evaluating the Efficacy, Safety and Immunogenicity of Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks of Angioedema in Patients With HAE
Brief Title: Efficacy, Safety and Immunogenicity Study of Recombinant Human C1 Inhibitor for the Treatment of Acute HAE Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C1 1310
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary Angioedema; HAE; Angioedema; Recombinant C1 Inhibitor; rhC1INH
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rhC1INH (Experimental)
  Interventions: Drug: rhC1INH
- Placebo (Saline) (Placebo Comparator)
  Interventions: Drug: Placebo (Saline)

INTERVENTIONS:
Drug: rhC1INH — One i.v. injection of rhC1INH at the dose of 50 U/kg, for patients up to 84 kg; one i.v. injection of rhC1INH at the dose of 4200U (2 vials) for patients of 84 kg body weight or greater.
  Arms: rhC1INH
Drug: Placebo (Saline) — One i.v. injection of saline (NaCl 0.9% w/v), equivalent in volume to the active treatment
  Arms: Placebo (Saline)

SUMMARY:
This study is being conducted to confirm the efficacy, safety, and immunogenicity of recombinant human C1 inhibitor (rhC1INH) at a dose of 50 U/kg when used for the treatment of acute angioedema attacks in Hereditary Angioedema (HAE) patients.

DETAILED DESCRIPTION:
HAE is characterized by recurrent localized angioedema caused by uncontrolled activation of the complement and contact systems due to a congenital deficiency of functional C1 inhibitor.

rhC1INH has been developed to offer a more widely available therapeutic alternative to the existing plasma-derived C1INH (pdC1INH) products that have been used in the treatment of acute angioedema attacks patients with HAE.

Patients who have qualified for enrollment in advance and who present to a study center within 5 hours of onset of an attack will be evaluated for eligibility. 75 eligible patients will be randomized (3:2) to receive an intravenous infusion of rhC1INH or saline in a double-blind fashion. Open-label rhC1INH may be provided as rescue medication to patients who do not experience the beginning of relief within 4 hours or who experience life-threatening oropharyngeal-laryngeal angioedema symptoms.

Any patient having received a randomized treatment will be allowed to receive treatment with rhC1INH in an open-label fashion for subsequent eligible attacks.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 13 years
* Signed written informed consent
* Clear clinical and laboratory diagnosis of HAE with baseline plasma level of functional C1INH of less than 50% of normal
* Willingness and ability to comply with all protocol procedures
* Clinical symptoms of an eligible HAE attack with onset less than 5 hours before the time of initial evaluation

Exclusion Criteria:

* Medical history of allergy to rabbits or rabbit-derived products (including rhC1INH), or positive anti-rabbit dander IgE test (cut off >0.35 kU/L; ImmunoCap® assay; Phadia or equivalent).
* A diagnosis of acquired C1INH deficiency (AAE)
* Pregnancy, or breastfeeding, or current intention to become pregnant
* Treatment with any investigational drug in the past 30 days
* Known or suspected addiction to drug and/or alcohol abuse
* Suspicion for an alternate explanation of the symptoms other than acute HAE attack

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (15):
  - Allergy, Asthma & Immunology, Assoc, Ltd., Scottsdale, Arizona
  - Allergy and Asthma Institute of the Valley, Granada Hills, California
  - UCLA Department of Medicine Division of Clinical Immunology, David Geffen School of Medicine, Los Angeles, California
  - USF Asthma, Allergy and Immunology Clinical Research Unit, Tampa, Florida
  - Family Allergy and Asthma Center, Atlanta, Georgia
  - Institute for Asthma and Allergy, P.C., Chevy Chase, Maryland
  - Asthma & Allergy Center - Washington University School of Medicine, St Louis, Missouri
  - University of Cincinnati Physicians, Inc., Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Baker Allergy, Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Pennsylvania State- Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
  - University of Texas - Medical Branch, Galveston, Texas
  - Allergy, Asthma & Immunology Clinic, P.A., Irving, Texas
  - Marycliff Allergy Specialists, Spokane, Washington
- UMHAT "Tsaritsa Yoanna - ISUL"; Clinic of Ear-Nose-Throat Diseases, Sofia, Bulgaria
- Ottawa Allergy Research Corp., Ottawa, Ontario, Canada
- Semmelweis University Faculty of Medicine, III Department of Internal Medicine, Budapest, Hungary
- Israel (2):
  - Allergy, Immunology & Angioedema Center,, Tel Litwinsky, Ramat Gan
  - Bnei-Zion Medical Centre, Clinical Immunology and Allergy Division, Haifa
- Ospedale Luigi Sacco, Azienda Ospedaliera - Polo Universitario II Divisione di Medicina Interna, Milan, Italy
- P.H.U. Clinic for Dermatology, Medical University Skopje, Unit of Allergology and Clinical Immunology, Skopje, North Macedonia
- Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Klinik Chorób Wewnętrznych, Poradnia Alergologiczna, Krakow, Poland
- Spitalul Clinic Judeţean Mureş Secţia Clinică Medicină Internă, Compartimentul de Alergologie şi Imunologie, Târgu Mureş, Romania
- Clinic for Immunology and Allergology, Belgrade, Serbia
- South Africa (2):
  - Allergy Diagnostic & Clinical Research Unit University of Cape Town Lung Institute, Mowbray
  - Wits Health Consortium (Pty) Ltd - Wits Donald Gordon Medical Centre, Parktown

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the double blind phase of the study, patients were randomized once to receive rhC1INH or Saline in a ratio of 3:2. After the randomized treatment, patiënts with subsequent attacks could be trated with open-label rhC1INH.
Pre-assignment Details: Patients could be enrolled into the open-label phase of the study after the initial randomized treatment.
Period: Double-blind Phase
Arm/Group | rhC1INH | Placebo (Saline)
Started | 44 | 31
Completed | 43 | 31
Not Completed | 1 | 0
Not completed — randomized not treated | 1 | 0
Period: Open Label Phase
Arm/Group | rhC1INH | Placebo (Saline)
Started | 24 (Not all Double-Blind Phase participants went on to Open Label Phase) | 20 (Not all Double Blind Phase participants went on to Open Label Phase)
Completed | 24 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhC1INH | Placebo (Saline) | Total
Number analyzed (Participants) | 44 | 31 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 42 | 29 | 71
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 19 | 47
  Male | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Time to Beginning of Relief of Symptoms
Description: Time to beginning of relief is the time lapsed from the beginning of the infusion of study medication to the beginning of a beneficial effect based on patient's responses to the Treatmetn Effect Questionnaire (TEQ) for the primary attack location. The beginning of relief is defined as the first timepoint at which
  * The patient reports any of the following answers for TEQ question 1: "A little better", "Better" or "Much better"; and;
  * The patient reports the following answer for TEQ question 2: "Yes"; and,
  * There is persistence in improvement at the next assessment time, i.e.either the same or a better response to Question 1 and "Yes" to Question 2.
Time Frame: Patients observed for 24 hours
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | rhC1INH | Placebo (Saline)
Number analyzed (Participants) | 43 | 31
minutes | 90 [61 to 150] | 152 [93 to NA] — The upper bound of the 95% confidence interval is not estimable due to censoring, and therefore an insufficient number of participants with events.

2. Secondary Outcome: Time to Minimal Symptoms
Description: The key secondary efficacy endpoint was the time to minimal symptoms at all locations. The time to achieving minimal symptoms was defined as an answer of "Yes" to TEQ question 3.
Time Frame: 24 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | rhC1INH | Placebo (Saline)
Number analyzed (Participants) | 44 | 31
minutes | 303 [240 to 720] | 483 [300 to 1440]

ADVERSE EVENTS:
Time Frame: From signing of the ICF till 90 days following each treated attack. If multiple attacks were treated, each was followed for 90 days.
Description: In the participants at risk rhC1INH arm group, patients that were randomized to Placebo in the Double Blind phase but received a rescue dose (rhC1INH) are included.
Arm/Group | rhC1INH | Placebo (Saline)
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/18
Other Adverse Events (participants affected / at risk) | 6/56 | 4/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhC1INH (N=56) | Placebo (Saline) (N=18)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhC1INH (N=56) | Placebo (Saline) (N=18)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibrin D-dimer increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To ensure against inadvertent disclosure of confidential information, the PI will provide Sponsor an opportunity to review any proposed publication/disclosure before it is submitted or otherwise disclosed. The PI will submit proposed manuscript, publication or disclosure to the Sponsor for comment at least 60 days prior to its submission/disclosure. If requested, the publishing party shall remove any Information (other than Study results) prior to submitting or disclosing the materials.